CLINICAL TRIAL: NCT04811131
Title: A Phase 2a, Proof of Concept, 24-Week, Parallel Group, Double Blind, Vehicle-Controlled Study of the Safety and Efficacy of ARQ-252 Cream 0.3% in Subjects With Non-Segmental Facial Vitiligo
Brief Title: Safety and Efficacy of ARQ-252 Cream 0.3% in Subjects With Non-Segmental Facial Vitiligo
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Arcutis Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARQ-252-213
Record Dates: First submitted 2021-03-18; First posted 2021-03-23 (Actual); Results first posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Intervention Model Description: This study is a parallel group, double blind, vehicle-controlled study in which subjects with non-segmental vitiligo will be randomized to ARQ-252 0.3% cream BID or vehicle cream BID, and active phototherapy or sham phototherapy for 24 weeks to affected areas of vitiligo on the face, neck, hands, forearms, and elbows, (Up to 15% total body BSA)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Active IP and Active Phototherapy (Active Comparator): ARQ-252 cream 0.3% BID with phototherapy.
  Interventions: Drug: ARQ-252 cream 0.3%; Device: NB-UVB phototherapy active treatment
- Active IP and Sham Phototherapy (Active Comparator): ARQ-252 cream 0.3% BID with sham phototherapy
  Interventions: Drug: ARQ-252 cream 0.3%; Device: NB-UVB phototherapy sham treatment
- Vehicle and Active Phototherapy (Placebo Comparator): ARQ-252 Vehicle cream BID with active phototherapy
  Interventions: Drug: ARQ-252 Vehicle cream; Device: NB-UVB phototherapy active treatment
- Vehicle and Sham Phototherapy (Placebo Comparator): ARQ-252 Vehicle cream BID with sham phototherapy
  Interventions: Drug: ARQ-252 Vehicle cream; Device: NB-UVB phototherapy sham treatment

INTERVENTIONS:
Drug: ARQ-252 cream 0.3% — ARQ-252 cream 0.3%
  Arms: Active IP and Active Phototherapy; Active IP and Sham Phototherapy
Drug: ARQ-252 Vehicle cream — ARQ-252 Vehicle cream
  Arms: Vehicle and Active Phototherapy; Vehicle and Sham Phototherapy
Device: NB-UVB phototherapy active treatment — NB-UVB phototherapy active treatment
  Arms: Active IP and Active Phototherapy; Vehicle and Active Phototherapy
Device: NB-UVB phototherapy sham treatment — NB-UVB phototherapy sham treatment
  Arms: Active IP and Sham Phototherapy; Vehicle and Sham Phototherapy

SUMMARY:
This study will assess the safety and efficacy of ARQ-252 cream in combination with NB-UVB phototherapy treatment in individuals with non-segmental facial vitiligo.

DETAILED DESCRIPTION:
This study is a Phase 2a, parallel group, double blind, vehicle-controlled study of the safety and efficacy of ARQ-252 0.3% cream in combination with NB-UVB phototherapy treatment in subjects with non-segmental facial vitiligo.

This study was prematurely terminated by the sponsor on 30-Jun-2021.

ELIGIBILITY:
Inclusion Criteria:

* Subject is legally competent to sign and give informed consent.
* Males and females ages 18 years and older (inclusive)
* Clinical diagnosis of non-segmental vitiligo involving face.
* A Facial Vitiligo Area Severity Index [F-VASI] score of ≥ 0.25 at baseline.
* Vitiligo of the face involving at least ≥ 0.25% body surface area (BSA) involvement (ie, one quarter of one handprint). Subjects may have non-facial vitiligo elsewhere which will not be included in the minimum BSA. The maximum BSA (total body inclusive of the face, whether or not in areas to be treated in this study) permitted is 15%.
* Subjects with vitiligo on the hands, forearms, or elbows agree to treat these areas in addition to the face, with investigational product and phototherapy.
* Subject agrees to discontinue all agents used to treat vitiligo from screening through the final safety follow-up visit. Over-the-counter preparations deemed acceptable by the Investigator and camouflage makeups are permitted.
* Female subject of childbearing potential (FOCBP) must have a negative serum pregnancy test at Screening and negative urine pregnancy test at Baseline (Visit 2). For FOCBP involved in any sexual intercourse that could lead to pregnancy: the subject must agree to use a highly effective contraceptive method for at least 4 weeks prior to Day 1. Additionally, from Day 1 until at least 4 weeks after the last investigational product administration, these subjects must agree to use at least 1 highly effective contraceptive method in addition to 1 barrier method.
* Female subject of non-childbearing potential must either be post-menopausal with spontaneous amenorrhea for at least 12 months prior to baseline (post-menopausal status will be confirmed with FSH testing) or have undergone surgical sterilization.
* Males, if engaging in sexual intercourse with a female who is pregnant or a female of child-bearing potential, must agree to use a condom every time during the study and every time subsequently until 4 weeks beyond the last dose of investigational product.
* Males must agree not to donate sperm from the first dose of investigational product until 4 weeks after the last dose of investigational product.
* Subject is in good health as judged by the Investigator, based on medical history, physical examination, 12-lead electrocardiogram (ECG), serum chemistry labs, hematology values, and urinalysis.

Exclusion Criteria:

* Subjects who have ever used skin bleaching treatments for treatment of vitiligo or other pigmented areas, eg, depigmenting agents such as monobenzyl ether of hydroquinone, including Benoquin® (Monobenzone)
* Use of any other prior and concomitant therapy that is a contraindication to phototherapy or may otherwise interfere with the objective of the study as per discretion of the Investigator, such as drugs that cause photosensitivity or skin pigmentation (eg, antibiotics such as tetracyclines, antifungals) within 8 weeks of Baseline (Visit 2).
* More than 33% leukotrichia in facial lesions (assessed via dermatoscope).
* Other forms of vitiligo (eg, segmental vitiligo); or other skin depigmentation disorder that would confound study assessments.
* Use of oral or systemic immunomodulating medications (eg, corticosteroids, azathioprine, methotrexate, cyclosporine) within 8 weeks of Baseline (Visit 2).
* Use of prescription or over-the-counter topical treatments that may affect vitiligo (eg, corticosteroids, tacrolimus/pimecrolimus, retinoids, vitamin D derivates, psoralens) within 4 weeks prior to Baseline (Visit 2).
* Use of any biological or experimental therapy for vitiligo within 24 weeks of Baseline (Visit 2) (or 5 half-lives, whichever is longer).
* Use of phototherapy (including laser and tanning beds) within 8 weeks prior to Baseline (Visit 2).
* Previous oral or topical JAK inhibitor therapy within 24 weeks prior to Baseline (Visit 2), and/or prior non-response to oral or topical JAK inhibitor therapy for vitiligo
* History of melanocyte-keratinocyte transplantation procedure (MKTP) or other surgical treatment for vitiligo.
* Contraindication to phototherapy, such as photosensitivity disorder (eg, lupus, polymorphic light eruption, solar urticaria, dermatomyositis) or use of photosensitizing or phototoxic medications.
* Subjects with clinically significant abnormal thyroid-stimulating hormone or free T4 at screening, or otherwise uncontrolled thyroid function at screening as determined by the investigator (Note: If the subject has a history of thyroid disease and is on treatment, the participant must be on a stable thyroid regimen for at least 3 months prior to baseline)
* History of chronic alcohol or drug abuse within 6 months prior to baseline.
* Subjects with a cytopenia at screening, defined as follows: Leukocytes < 3 × 10^9/L (2.5 × 10^9/L for subjects who are African-American), Neutrophils < lower limit of normal (<1.5x10^9/L), Lymphocytes < 0.8 × 10^9/L, Hemoglobin < 10 g/dL, Platelets < 100 × 10^9/L.
* Subjects with current or a history of non-skin cancer within 5 years with the exception carcinoma in situ of the cervix.
* Subjects with greater than 3 adequately treated nonmetastatic basal cell carcinomas (BCC) or squamous cell carcinomas (SCC) within 12 months prior to Baseline (Visit 2), or a previous history of multiple BCC or SCC on any area of the body, which may pose additional risks from participation in the study, in the opinion of the Investigator.
* Subjects with previous history of melanoma anywhere on the body, or basal cell carcinoma (BCC), squamous cell carcinoma (SCC), or actinic keratosis (AK) on the face, neck, hands, forearms, or elbows.
* Subjects that have received live vaccine therapy less than 4 weeks prior Baseline (Visit 2), or anticipate receiving a live or live-attenuated vaccination during the course of the study, have received immunosuppressive drugs less than 4 weeks prior Baseline, or have known infection with mycobacterium tuberculosis, hepatitis B or C, or HIV, or have a diagnosis of an immunodeficiency disorder.
* Subject had a major surgery within 4 weeks prior to Baseline or has a major surgery planned during the study.
* Subjects with severe renal insufficiency (as evidenced by estimated glomerular filtration rate <40 mL/min) or with severely impaired liver function (Child-Pugh Class C), ALT or AST ≥ 2 × ULN, total bilirubin > 1.5 x ULN, or total bilirubin > ULN and ≤ 1.5 x ULN AND direct bilirubin is > 35% of total bilirubin, ALP ≥ 2x ULN
* Subjects with known or suspected hypersensitivity to component(s) of the investigational product.
* Pregnant or lactating women or women planning to become pregnant during the study and / or within 28 days following the last dose of investigational product.
* Subjects who cannot discontinue the use of strong systemic Cytochrome P-450 CYP3A4 inducers e.g., efavirenz, nevirapine, glucocorticoids, barbiturates (including phenobarbital), phenytoin, rifampin and carbamazepine for 2 weeks prior to Baseline and during the study period.
* Subjects who cannot discontinue the use of strong systemic Cytochrome P-450 CYP3A4 inhibitors e.g., indinavir, nelfinavir, ritonavir, clarithromycin, itraconazole, ketoconazole, fluconazole, nefazodone, saquinavir, suboxone and telithromycin for 2 weeks prior to Baseline and during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2021-03-04 (Actual); Primary Completion 2021-08-09 (Actual); Study Completion 2021-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Berk, MD, Study Director — Arcutis Biotherapeutics, Inc.
Locations (5):
- United States (5):
  - Arcutis Site 123, San Diego, California
  - Arcutis Site 167, Coral Gables, Florida
  - Arcutis Clinical Site 102, Rolling Meadows, Illinois
  - Arcutis Site 162, Austin, Texas
  - Arcutis Clinical Site 163, Pflugerville, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomized at 31 study centers in the United States and Canada.
Pre-assignment Details: The study was early terminated and only available descriptive statistics are shown.
Groups:
- Active IP and Active Phototherapy: Participants receive ARQ-252 cream 0.3% twice daily (BID) with phototherapy for 24 weeks.
- Active IP and Sham Phototherapy: Participants receive ARQ-252 cream 0.3% BID with sham phototherapy for 24 weeks.
- Vehicle and Active Phototherapy: Participants receive vehicle cream BID with phototherapy for 24 weeks.
- Vehicle and Sham Phototherapy: Participants receive vehicle cream BID with sham phototherapy for 24 weeks.
Period: Overall Study
Arm/Group | Active IP and Active Phototherapy | Active IP and Sham Phototherapy | Vehicle and Active Phototherapy | Vehicle and Sham Phototherapy
Started | 34 | 37 | 31 | 12
Completed | 0 | 0 | 0 | 0
Not Completed | 34 | 37 | 31 | 12
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Sponsor request | 31 | 35 | 27 | 10
Not completed — Withdrawal by Subject | 3 | 1 | 3 | 1

BASELINE CHARACTERISTICS:
Population: The Baseline Analysis Population is based on all treated participants.
Groups:
- Active IP and Active Phototherapy: Participants receive ARQ-252 cream 0.3% BID with phototherapy.
- Active IP and Sham Phototherapy: Participants receive ARQ-252 cream 0.3% BID with sham phototherapy.
- Vehicle and Active Phototherapy: Participants receive vehicle cream BID with phototherapy.
- Vehicle and Sham Phototherapy: Participants receive vehicle cream BID with sham phototherapy.
- Total: Total of all reporting groups
Arm/Group | Active IP and Active Phototherapy | Active IP and Sham Phototherapy | Vehicle and Active Phototherapy | Vehicle and Sham Phototherapy | Total
Number analyzed (Participants) | 34 | 36 | 30 | 12 | 112
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.5 (12.75) | 46.2 (10.84) | 47.9 (12.90) | 43.5 (7.23) | 46.8 (11.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 20 | 8 | 7 | 53
  Male | 16 | 16 | 22 | 5 | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 9 | 10 | 4 | 35
  Not Hispanic or Latino | 22 | 26 | 20 | 8 | 76
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American-Indian or Alaska Native | 1 | 0 | 3 | 2 | 6
  Asian | 4 | 4 | 1 | 1 | 10
  Black or African American | 1 | 5 | 3 | 0 | 9
  White | 26 | 27 | 21 | 7 | 81
  Other | 2 | 0 | 1 | 2 | 5
  More than One Race | 0 | 0 | 1 | 0 | 1
Facial Vitiligo Area Scoring Index (F-VASI) Baseline Score [Mean (Standard Deviation); unit: units on a scale] — F-VASI measures the % of vitiligo involvement (percentage of body surface area [BSA]) and the degree of depigmentation: 0% (none), 10% (only specks), 25% (pigmented area > depigmented area), 50% (depigmented and pigmented areas equal), 75% (depigmented area > pigmented area), 90% (specks of pigment), or 100% (no pigment). F-VASI was then derived by multiplying the values assessed for the vitiligo involvement by the percentage of affected skin for each site on the face and summing the values of all sites (possible range: 0-3; lower scores indicate increased improvement).
  units on a scale | 0.743 (0.5970) | 0.820 (0.8062) | 0.656 (0.5943) | 1.061 (0.6571) | 0.779 (0.6780)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving 75% Reduction in Facial Vitiligo Area Scoring Index (F-VASI) Score (F-VASI75) at Week 24
Description: Achievement of F-VASI75 was declared with a ≥75% improvement from Baseline in F-VASI. F-VASI measures the % of vitiligo involvement (percentage of body surface area [BSA]) and the degree of depigmentation: 0% (none), 10% (only specks), 25% (pigmented area > depigmented area), 50% (depigmented and pigmented areas equal), 75% (depigmented area > pigmented area), 90% (specks of pigment), or 100% (no pigment). F-VASI was then derived by multiplying the values assessed for the vitiligo involvement by the percentage of affected skin for each site on the face and summing the values of all sites (possible range: 0-3; lower scores indicate increased improvement).
Time Frame: Week 24
Population: No participants were analyzed due to early study termination.
Groups:
- Active IP and Active Phototherapy: Participants receive ARQ-252 cream 0.3% BID with phototherapy for 24 weeks.
Arm/Group | Active IP and Active Phototherapy | Active IP and Sham Phototherapy | Vehicle and Active Phototherapy | Vehicle and Sham Phototherapy
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Secondary Outcome: Percentage of Change From Baseline in F-VASI Score
Description: The mean (SD) percentage change from baseline in F-VASI scores across study time points is presented. F-VASI measures the % of vitiligo involvement (percentage of body surface area [BSA]) and the degree of depigmentation: 0% (none), 10% (only specks), 25% (pigmented area > depigmented area), 50% (depigmented and pigmented areas equal), 75% (depigmented area > pigmented area), 90% (specks of pigment), or 100% (no pigment). F-VASI was then derived by multiplying the values assessed for the vitiligo involvement by the percentage of affected skin for each site on the face and summing the values of all sites (possible range: 0-3; lower scores indicate increased improvement).
Time Frame: Weeks 4, 8, 12, 16, 20, and 24
Population: All randomized participants with data available are included.
Measure: Mean (Standard Deviation); unit: percentage of change from baseline
Arm/Group | Active IP and Active Phototherapy | Active IP and Sham Phototherapy | Vehicle and Active Phototherapy | Vehicle and Sham Phototherapy
Number analyzed (Participants) | 34 | 37 | 31 | 12
percentage of change from baseline
  Week 4: number analyzed (Participants) | 18 | 16 | 15 | 5
  Week 4 | -21.009 (25.0121) | -7.775 (11.8841) | -11.589 (21.5439) | 2.857 (6.3888)
  Week 8: number analyzed (Participants) | 8 | 7 | 6 | 2
  Week 8 | -57.160 (27.3703) | -27.917 (23.4974) | -39.570 (27.5064) | -16.667 (23.5702)
  Week 12: number analyzed (Participants) | 1 | 6 | 1 | 0
  Week 12 | -62.963 (NA) — NA due to n=1 | -54.157 (16.7882) | -33.333 (NA) — NA due to n=1 |
  Week 16: number analyzed (Participants) | 0 | 2 | 0 | 0
  Week 16 |  | -10.100 (55.6893) |  |
  Week 20: number analyzed (Participants) | 0 | 0 | 0 | 0
  Week 24: number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Change From Baseline in Facial Body Surface Area (F-BSA) Score
Description: The change from baseline in F-BSA affected over time. The endpoint was not assessed due to early study termination.
Time Frame: Weeks 4, 8, 12, 16, 20, and 24
Population: No participants were analyzed due to early study termination.
Arm/Group | Active IP and Active Phototherapy | Active IP and Sham Phototherapy | Vehicle and Active Phototherapy | Vehicle and Sham Phototherapy
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: Change From Baseline in Vitiligo Noticeability Scale (VNS) Score
Description: The VNS is a patient-reported measure of vitiligo treatment success, which has a 5-point scale, with 1 being more noticeable and 5 being no longer noticeable. The VNS will be completed for vitiligo on the face. The endpoint was not assessed due to early study termination.
Time Frame: Weeks 4, 8, 12, 16, 20, and 24.
Population: No participants were analyzed due to early study termination.
Arm/Group | Active IP and Active Phototherapy | Active IP and Sham Phototherapy | Vehicle and Active Phototherapy | Vehicle and Sham Phototherapy
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Change From Baseline in Vitiligo Quality of Life (VitiQOL)
Description: Change from Baseline in the VitiQoL, an instrument consisting of 16-item questionnaire (with a 7-point numerical scale from 0 - Not at all to 6 - All of the time) designed to assess disease specific health-related quality of life (HRQL) in patients suffering from vitiligo and also provide an objective measure of disease status, burden of disease, and treatment outcome. The endpoint was not assessed due to early study termination.
Time Frame: Weeks 4, 8, 12, 16, 20, and 24
Population: No participants were analyzed due to early study termination.
Arm/Group | Active IP and Active Phototherapy | Active IP and Sham Phototherapy | Vehicle and Active Phototherapy | Vehicle and Sham Phototherapy
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: Change From Baseline in Patient Global Impression of Change-Vitiligo (PaGIC-V)
Description: The PaGIC-V category, a 7-point scale comparing facial vitiligo at baseline with the subject's treated facial vitiligo at the study visit (with 1- very much improved and 7 - very much worse), and time to achieve a PaGIC-V of very much improved or much improved. The endpoint was not assessed due to early study termination.
Time Frame: Week 4, 8, 12, 16, 20, and 24
Population: No participants were analyzed due to early study termination.
Arm/Group | Active IP and Active Phototherapy | Active IP and Sham Phototherapy | Vehicle and Active Phototherapy | Vehicle and Sham Phototherapy
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: Percentage of Participants Achieving 50% Reduction in F-VASI Score (F-VASI50)
Description: The percentage of participants achieving F-VASI50. The endpoint was not assessed due to early study termination.
Time Frame: Week 4, 8, 12, 16, 20, and 24
Population: No participants were analyzed due to early study termination.
Arm/Group | Active IP and Active Phototherapy | Active IP and Sham Phototherapy | Vehicle and Active Phototherapy | Vehicle and Sham Phototherapy
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Secondary Outcome: Time to Achieve F-VASI50
Description: The time to achieve F-VASI50. The endpoint was not assessed due to early study termination.
Time Frame: Week 4, 8, 12, 16, 20, and 24
Population: No participants were analyzed due to early study termination.
Arm/Group | Active IP and Active Phototherapy | Active IP and Sham Phototherapy | Vehicle and Active Phototherapy | Vehicle and Sham Phototherapy
Number analyzed (Participants) | 0 | 0 | 0 | 0

9. Secondary Outcome: Percentage of Participants Achieving 90% Reduction in F-VASI Score (F-VASI90)
Description: The percentage of participants achieving F-VASI90. The endpoint was not assessed due to early study termination.
Time Frame: Week 4, 8, 12, 16, 20, and 24
Population: No participants were analyzed due to early study termination.
Arm/Group | Active IP and Active Phototherapy | Active IP and Sham Phototherapy | Vehicle and Active Phototherapy | Vehicle and Sham Phototherapy
Number analyzed (Participants) | 0 | 0 | 0 | 0

10. Secondary Outcome: Achievement of Success in Facial Static Investigator Global Assessment (FsIGA)
Description: The percentage of subjects with FsIGA, (a four point scale of vitiligo severity for the face only) of clear or almost clear (0 or 1) and time to achieve FsIGA of clear or almost clear (0 or 1). The endpoint was not assessed due to early study termination.
Time Frame: Week 4, 8, 12, 16, 20, and 24
Population: No participants were analyzed due to early study termination.
Groups:
- Vehicle and Sham Phototherapy: Participants receive vehicle cream with sham phototherapy for 24 weeks.
Arm/Group | Active IP and Active Phototherapy | Active IP and Sham Phototherapy | Vehicle and Active Phototherapy | Vehicle and Sham Phototherapy
Number analyzed (Participants) | 0 | 0 | 0 | 0

11. Secondary Outcome: Time to Achieve F-VASI75
Description: The time to achieve F-VASI75 50. The endpoint was not assessed due to early study termination.
Time Frame: Week 4, 8, 12, 16, 20, and 24
Population: No participants were analyzed due to early study termination.
Arm/Group | Active IP and Active Phototherapy | Active IP and Sham Phototherapy | Vehicle and Active Phototherapy | Vehicle and Sham Phototherapy
Number analyzed (Participants) | 0 | 0 | 0 | 0

12. Secondary Outcome: Achievement of Success in FsIGA Score
Description: FsIGA of clear or almost clear (0 or 1) plus 2-grade improvement from baseline. The endpoint was not assessed due to early study termination.
Time Frame: Week 4, 8, 12, 16, 20, and 24
Population: No participants were analyzed due to early study termination.
Arm/Group | Active IP and Active Phototherapy | Active IP and Sham Phototherapy | Vehicle and Active Phototherapy | Vehicle and Sham Phototherapy
Number analyzed (Participants) | 0 | 0 | 0 | 0

13. Secondary Outcome: Time to PaGIC-V Score of Very Much Improved or Improved
Description: The time to a PaGIC-V score of 1 'very much improved' or 2 'improved'. The PaGIC-V category, a 7-point scale comparing facial vitiligo at baseline with the subject's treated facial vitiligo at the study visit (with 1- very much improved and 7 - very much worse), and time to achieve a PaGIC-V of very much improved or much improved. The endpoint was not assessed due to early study termination.
Time Frame: Week 4, 8, 12, 16, 20, and 24
Population: No participants were analyzed due to early study termination.
Arm/Group | Active IP and Active Phototherapy | Active IP and Sham Phototherapy | Vehicle and Active Phototherapy | Vehicle and Sham Phototherapy
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to ~22 weeks
Description: All treated participants are included
Groups:
- Vehicle and Active Phototherapy: Participants receive vehicle cream BID h phototherapy for 24 weeks.
Arm/Group | Active IP and Active Phototherapy | Active IP and Sham Phototherapy | Vehicle and Active Phototherapy | Vehicle and Sham Phototherapy
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/36 | 0/30 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/36 | 0/30 | 0/12
Other Adverse Events (participants affected / at risk) | 4/34 | 1/36 | 3/30 | 5/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Active IP and Active Phototherapy (N=34) | Active IP and Sham Phototherapy (N=36) | Vehicle and Active Phototherapy (N=30) | Vehicle and Sham Phototherapy (N=12)
Oral herpes (Infections and infestations) | 0 | 0 | 2 | 0
Sunburn (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Dysguesia (Nervous system disorders) | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Application site pain (General disorders) | 2 | 1 | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-04-14): https://cdn.clinicaltrials.gov/large-docs/31/NCT04811131/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-28): https://cdn.clinicaltrials.gov/large-docs/31/NCT04811131/SAP_001.pdf